CLINICAL TRIAL: NCT01728103
Title: Prospective Collection of Female First-catch Urine, Vaginal Swab,Cervical, and Endocervical Swab Specimens for Testing With the APTIMA Assays
Brief Title: Prospective Collection of Female Specimens for Testing With Gen-Probe APTIMA (Registered Trademark) Assays
Status: Terminated | Type: Observational
Why Stopped: Corporate decision to spend money on other development programs.
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: ATVTS-US12-001; AC2PS-US12-002 (Other: Gen-Probe); ATVPS-US12-001 (Other: Gen-Probe); ATVTS-US12-003 (Other: Gen-Probe)
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Chlamydia Infections; Gonorrhea; Trichomonas Infections
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Trichomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine; endocervical and vaginal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment
  Interventions: Device: APTIMA® Trichomonas vaginalis & APTIMA® COMBO 2® Assays

INTERVENTIONS:
Device: APTIMA® Trichomonas vaginalis & APTIMA® COMBO 2® Assays — In Vitro Diagnostic Assays

SUMMARY:
The objective of this study is to obtain female first-catch urine, vaginal, cervical and endocervical swabs for testing with multiple APTIMA Assays on the Gen-Probe PANTHER® and TIGRIS® Systems.

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 16 years of age at the time of enrollment and is currently sexually active (has had penile/vaginal intercourse within the past 12 months)
* The subject and/or legally authorized representative is willing to undergo the informed consent process prior to study participation (a minor will need the documented consent of his/her parent or legal guardian, unless the site has an institutional review board [IRB]-approved waiver for parental consent for minors)

In addition, the subject must meet at least one of the following criteria:

* The subject reports symptoms consistent with a suspected sexually transmissible infection (STI) such as abnormal discharge, genital itching, pain/discomfort during sexual intercourse or urination, and/or lower abdominal discomfort
* Subject is asymptomatic and known to be partners with, or a contact of, a person with a confirmed or suspected STI(s)
* Subject is asymptomatic and undergoing screening evaluation for possible STIs
* Subject is asymptomatic and undergoing a routine examination with a pelvic examination

Exclusion Criteria:

* The subject took antibiotic medications within the last 21 days
* Subject already participated in this study
* Subject has a history of illness that the principal investigator (PI) or designee considers could interfere with or affect the conduct, results, and/or completion of the clinical trial
* Subject has a history of illness that the PI or designee considers could create an unacceptable risk to the subject if enrolled

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Female subjects at least 16 years of age, with or without symptoms of sexually transmitted disease.
Sampling Method: Probability Sample
Enrollment: 1336 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Qualitative detection of ribosomal RNA from Chlamydia trachomatis and/or Neisseria gonorrhoeae (NG) and Trichomonas vaginalis (TV) to aid in the diagnosis of chlamydial and/or gonococcal and/or trichomonal urogenital disease | approximately one year

CONTACTS AND LOCATIONS:
Overall Officials: Renee Wait, Study Director — Gen-Probe, Incorporated
Locations (14):
- United States (14):
  - Infectious Diseases STD Program University of Alabama at Birmingham, Birmingham, Alabama
  - Medical Center for Clinical Research, San Diego, California
  - Healthcare Clinical Data, North Miami, Florida
  - Mount Vernon Clinical Research, Sandy Springs, Georgia
  - Louisiana State University Health Sciences Center Dept. of Medicine, Infectious Disease, New Orleans, Louisiana
  - John Hopkins University, Baltimore, Maryland
  - New England Center for Clinical Research, Fall River, Massachusetts
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center Division of Pediatric & Adolescent Gynecology, Cincinnati, Ohio
  - Planned Parenthood Southeastern Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Jackson Clinic, Jackson, Tennessee
  - Planned Parenthood Gulf Coast, Houston, Texas
  - Tidewater Clinical Research, Norfolk, Virginia